CLINICAL TRIAL: NCT05685706
Title: Knee-Hip-Spine Harmony: The Relationship Between Sagittal Spinal Alignment in Total Hip/Knee Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH110-REC2-030
Record Dates: First submitted 2022-12-29; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Cases Who Received TKA/THA
Keywords: Total hip/knee arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Concomitant osteoarthritis of hip/knee joint and lumbar spinal degeneration is commonly seen in elderly population. These degeneration changes of spine would change sagittal or coronal alignment and spinal flexibility in varies degrees. Total hip and knee arthroplasty (THA/TKA) are among the most successful orthopedic operations performed, aiming at the alleviation of osteoarthritic pain. Normal alignment of the spine and pelvis in the sagittal plane is critical to maintain an upright standing position with minimal energy consumption. However, there is a scarcity of studies on how THA or TKA influences the parameters of the spine and the pelvis.

Compared with the balance of coronal plane, more attention is paid to the balance of sagittal plane. The objectives of this study are to investigate changes in the truncal parameters after THA or TKA and assess whether these parameters are improved or deteriorated after these operations.

ELIGIBILITY:
Inclusion Criteria:

1. Primary degenerative arthritis of the knee or hip
2. Those who have undergone artificial knee or hip replacement surgery
3. Follow up surgery for at least 1 year
4. Track the whole trunk lower limb sagittal plane coronal aligament before and after surgery

Exclusion Criteria:

1. Previous hip surgery
2. Previous spine surgery
3. Contracture after hip fusion surgery
4. Scoliosis over 10 degrees combined with neuropathy
5. Patients with flexion contracture after knee joint surgery
6. Rheumatoid arthritis lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Concomitant osteoarthritis of hip/knee joint and lumbar spinal degeneration patients who take Total hip and knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
The Forgotten Joint Score-12 (FJS-12) | Post-operative at 24th month
  The Forgotten Joint Score-12 (FJS-12) is a validated patient-reported outcome measure (PROM) tool designed to assess artificial prosthesis awareness during daily activities following total hip arthroplasty (THA). The Forgotten Joint Score consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities (Rosinsky et al., 2019).
EQ-5D | Post-operative at 24th month
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan